CLINICAL TRIAL: NCT06497764
Title: A Pilot, Randomized, Non-blinded, Single-center Study of the Efficacy of a Vibrational Anesthesia (VA) Device on Reducing Pain During Platelet Rich Plasma (PRP) Scalp Treatment for Alopecia
Brief Title: Evaluating Vibrational Anesthesia in Scalp Platelet Rich Plasma (PRP)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Departmental research administration decided to close the study as there had been no enrollment. No participants were screened or consented.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-00472
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

ARMS (2):
- Control (PRP Alone), then Intervention (PRP with VA) (Experimental): Participants in this study arm will receive treatment with PRP alone first, then PRP+VA second. The first half of the scalp of each patient will be randomized to receive standard-of-care PRP alone. The second half of the scalp of each patient will receive VA via a device during the standard-of-care PRP treatment.
  Interventions: Device: Vibrational Anesthesia (VA) Device; Procedure: PRP Treatment
- Intervention (PRP with VA), then Control (PRP Alone) (Experimental): Participants in this study arm will receive treatment with PRP+VA first, then PRP alone second. The first half of the scalp of each patient will be randomized to receive VA via a device during the standard-of-care PRP treatment.. The second half of the scalp of each patient will receive standard-of-care PRP treatment alone.
  Interventions: Device: Vibrational Anesthesia (VA) Device; Procedure: PRP Treatment

INTERVENTIONS:
Device: Vibrational Anesthesia (VA) Device — The half of the patient's scalp randomized to receive VA during PRP treatment will receive VA via the Buzzy bee-striped personal. The device is powered by two AAA batteries and is indicated for use for pain reduction. It uses the Melzack and Wall's Gait Control theory, which states that activation of non-nociceptive fibers can interfere with signals from pain fibers to inhibit overall sensation of pain.
  Other Names: Buzzy bee-striped personal
Procedure: PRP Treatment — PRP (a needle-related procedure) will be delivered per routine standard of care.

SUMMARY:
This study is prospective, single-site, randomized split-scalp pilot and survey study of patients at the NYU Skin and Cancer Clinic or the Faculty Group Practice. The investigators will randomize half of the scalp of each patient: one half will receive vibrational anesthesia (VA) via a device and the other half will not. Approximately 100 unique patients will be recruited (there will only be one study group). During the standard of care platelet rich plasma (PRP) procedure, a REDCap survey questionnaire will be provided asking the patients to rate their pain with the visual analogue scale (VAS). A simple paired t-test will be used to test significant improvement in pain scores between the two halves of the scalp.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received at least one treatment of PRP to the scalp, which may include the PRP procedure performed day of.
* Able to participate in study procedures.
* Able to provide consent.

Exclusion Criteria:

* Patients missing the following data will be excluded from the final analysis: Patient age, gender, type of alopecia, PRP documentation.
* Patients unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Rating of Pain Perception at End of Procedure | End of procedure (About 10 minutes, Day 1)
  At the end of the 10-minute PRP procedure, participants will rate their pain on: 1) The side of the scalp with no VA, and 2) the side of the scalp with VA. Participants will rate pain using a VAS, where pain is rated on a 0-10 scale; larger values indicate greater pain levels.

SECONDARY OUTCOMES:
Percentage of Participants who Opt to use VA among Participants in the "Control, then Intervention" Arm | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Lo Sicco, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to Dr. Kristen Lo Sicco. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Kristen.losicco@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.